CLINICAL TRIAL: NCT04907032
Title: Title: A Randomized Clinical Trial Comparing Percutaneous Tibial Nerve Stimulation in Combination With Mirabegron to Percutaneous Tibial Nerve Stimulation Plus Placebo in Women With Refractory OAB Symptoms
Brief Title: Posterior Tibial Nerve Stimulation (PTNS) Plus Mirabegron to Treat Refractory OAB Symptoms (PTNS-M Study)
Acronym: PTNS-M
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Russell Stanley, DO, Instructor Fellow, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300006806-001
Record Dates: First submitted 2021-05-18; First posted 2021-05-28 (Actual); Results first posted 2023-07-20 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-06

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — mirabegron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Posterior Tibial Nerve Stimulation with Mirabegron (Experimental): One arm of the study will receive PTNS combined with mirabegron. In the PTNS with mirabegron arm, the patient will take a 50 mg dose daily for 12 weeks of the trial. This arm of the study will have 27 patients randomized to this arm of the study. The percutaneous approach entails insertion of a 36-gauge needle electrode at a 60 degree angle approximately 5 cm or 3 finger breadths cephalad to the medial malleolus and posterior to the tibia. A portable electrical stimulator delivers an adjustable current in the range of 0.5-9 mA. The generators commonly are set for a pulse frequency of 20 Hz with a goal of creating a motor and/or sensory response in the foot. The stimulation sessions last for 30 min once per week for 12 continuous weeks.
  Interventions: Drug: Mirabegron 50 MG; Device: Posterior Tibial Nerve Stimulation (PTNS)
- Posterior Tibial Nerve Stimulation Plus Placebo (Placebo Comparator): The other arm of the study will receive PTNS with placebo. In the PTNS with placebo arm, the patient will receive a placebo daily during the 12-week trial. PTNS will be performed as described: The percutaneous approach entails insertion of a 36-gauge needle electrode at a 60 degree angle approximately 5 cm or 3 finger breadths cephalad to the medial malleolus and posterior to the tibia. A portable electrical stimulator delivers an adjustable current in the range of 0.5-9 mA. The generators commonly are set for a pulse frequency of 20 Hz with a goal of creating a motor and/or sensory response in the foot. The stimulation sessions last for 30 min once per week for 12 continuous weeks.
  Interventions: Device: Posterior Tibial Nerve Stimulation (PTNS)

INTERVENTIONS:
Drug: Mirabegron 50 MG — Posterior Tibial Nerve Stimulation with Mirabegron vs. Posterior Tibial Nerve Stimulation Plus Placebo
  Other Names: Posterior Tibial Nerve Stimulation (PTNS)
  Arms: Posterior Tibial Nerve Stimulation with Mirabegron
Device: Posterior Tibial Nerve Stimulation (PTNS) — Posterior Tibial Nerve Stimulation with Mirabegron vs. Posterior Tibial Nerve Stimulation Plus Placebo

SUMMARY:
Abstract

Introduction: Urgency Urinary Incontinence (UUI) is a common condition with a prevalence of 9-31% in women in the United States. Despite current treatments, a high number of women have symptoms refractory to first- and second-line treatment approaches.

Aims: The primary aim of this randomized controlled trial is to compare the efficacy of percutaneous tibial nerve stimulation (PTNS) and mirabegron treatment versus PTNS with placebo on change in the number of UUI episodes over a 12-week treatment course. Secondary aims include comparing the efficacy of combined treatment of PTNS and mirabegron versus PTNS with placebo on improvement in urinary incontinence symptom specific distress and quality of life related to UUI over a 12-week course of PTNS.

Methods: A total of 54 consented participants will be recruited and randomized with 27 patients in the PTNS with mirabegron (daily 50 mg dose for the 12-week course) group and 27 patients in the PTNS with placebo group. Demographics and baseline data will be analyzed by student's t-test and chi-squared test or Fischer's Exact test as appropriate.

Hypothesis: We anticipate that combination therapy will prove superior to monotherapy for reducing the number of UUI episodes over a 12-week treatment course.

DETAILED DESCRIPTION:
Specific Aims:

Introduction/Background: Urgency Urinary Incontinence (UUI) remains a challenging clinical problem for urogynecologists as they treat women and seek to find better therapies. There is a wealth of literature addressing individual therapies for first, second, and third line treatments for UUI. There are three main third line treatment options for UUI including percutaneous tibial nerve stimulation (PTNS), sacral neuromodulation, and intradetrusor botox. At the current time, there are limited studies that have looked at a combination of second and third-line therapy therapies for UUI. While some anticholinergic medications have been studied in combination with percutaneous tibial nerve stimulation (PTNS) such as solifenacin, tolterodine, and trospium, there is limited data on the combination of mirabegron, a beta-3 agonist, and PTNS for treatment of refractory UUI. The studies that looked at anticholinergic medications in combination with PTNS revealed improvement in UUI compared to PTNS plus placebo. However, there are patients who do not tolerate anticholinergic medications well because of side effects. A relatively new finding as reported by the American Urogynecologic Society (AUGS) about avoiding anticholinergic medications in women greater than age 70 secondary to increased risk for cognitive impairment, dementia, and Alzheimer's disease is further impetus to conduct this trial [1]. The rationale for studying mirabegron in combination with PTNS versus PTNS plus placebo is important as mirabegron does not have the significant side effect profile that anticholinergic medications have and better tolerated in the older population. Therefore, more research should be performed to evaluate the effect of the combination of mirabegron and PTNS for refractory UUI. The purpose of this study is to evaluate the combination of PTNS and mirabegron and compare that to PTNS plus placebo in the treatment of refractory UUI.

Hypothesis: Combination therapy of PTNS and mirabegron, a beta-3 agonist, will contribute to greater improvement in the number of urgency urinary incontinence episodes as measured by a 3-day bladder diary compared to PTNS plus placebo in women.

Method: This is a randomized clinical trial comparing the efficacy of combination therapy with PTNS plus mirabegron to PTNS plus placebo in women with refractory urgency urinary incontinence.

Primary Aim: The primary aim of this study is to compare the efficacy of combined treatment of PTNS and mirabegron versus PTNS plus placebo on change in the number of UUI episodes at 12 weeks.

Secondary Aims:

* Comparing urinary symptom specific distress and quality of life over a 12-week course of PTNS.
* Comparing the side effect/adverse event profile of combined treatment of PTNS and mirabegron versus PTNS plus placebo over a 12-week course of PTNS
* Comparing the treatment efficacy and adverse events of combined treatment of PTNS and mirabegron versus PTNS plus placebo in women > 70 years of age as a sub analysis within the study

ELIGIBILITY:
Inclusion Criteria:

* Female patients > 18 years old at UAB facilities with refractory urgency urinary incontinence that have failed first line and second line treatments
* Ability to consent
* Ability to complete all study related items and interviews

Exclusion Criteria:

* Patients with a history of any known or determined urinary retention or urinary tract obstruction
* PVR > 150 ml in clinic prior to the start of PTNS
* History of bladder augmentation surgery
* Patients who are pregnant or who have the suspicion of pregnancy
* Uncontrolled hypertension
* Hypersensitivity to mirabegron
* Superficial and/or deep skin infection where PTNS intervention is required
* Spinal cord injury or clinically significant neurological disorders known to affect urgency urinary incontinence
* Bleeding diathesis
* Failure of previous third line treatment options such as sacral neuromodulation, PTNS, or Botox
* Pacemaker, implantable defibrillator
* Current use of Interstim sacral nerve stimulator or TENS in the pelvic region, back, or legs
* Coagulopathy
* Chronic swollen, infected, inflamed skin or skin eruptions (e.g., phlebitis, thrombophlebitis, varicose veins) in the region where the PTNS needles or surface electrodes would be placed
* Metal implant in foot/toes near TENS electrode location
* Marked sensory deficit (numbness) of feet or ankles in the region where the PTNS needles or surface electrodes would be placed
* Currently pregnant or planning to become pregnant during the course of the study
* Unwilling to use acceptable form of contraceptive if the participant is of childbearing potential
* Unable or unwilling to complete the 3-day bladder diary
* Visual impairment prohibiting reading the paper diary
* Inability to provide informed consent, complete questionnaires independently, or to attend intervention sessions
* Unable to speak, read, or write in English

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2023-04-01 (Actual); Study Completion 2023-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Russell F Stanley, DO, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: October 2021 to April 2023
Pre-assignment Details: 54 subjects were randomized and participated in the informed consent process. 7 subjects in the mirabegron plus posterior tibial nerve stimulation arm did not complete the study because they did not comply with showing up for all 12 study visits. There was 1 subject in the placebo to match plus posterior tibial nerve stimulation group who did not complete the study for the same reason.
Period: Overall Study
Arm/Group | Posterior Tibial Nerve Stimulation With Mirabegron | Posterior Tibial Nerve Stimulation Plus Placebo
Started | 27 | 27
Completed (withdrew because could not complete 12-week PTNS protocol.) | 20 | 26 (withdrew because could not complete 12-week PTNS protocol.)
Not Completed | 7 | 1
Not completed — Withdrawal by Subject | 7 | 1

BASELINE CHARACTERISTICS:
Population: Ch-squared tests or Fischer's exact tests were used to measure categorical variables
Groups:
- Total: Total of all reporting groups
Arm/Group | Posterior Tibial Nerve Stimulation With Mirabegron | Posterior Tibial Nerve Stimulation Plus Placebo | Total
Number analyzed (Participants) | 27 | 27 | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 18 | 39
  >=65 years | 6 | 9 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.8 (16.7) | 56.6 (14.7) | 56.2 (15.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 27 | 54
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 13 | 26
  White | 14 | 14 | 28
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African | 13 | 13 | 26
  White | 14 | 14 | 28
Region of Enrollment [Number; unit: participants]
  United States | 27 | 27 | 54

OUTCOME MEASURES:

1. Primary Outcome: Change in the Number of UUI Episodes Over a 3-day Voiding Diary Pre- vs. Post-treatment. This Includes a Baseline Measure Pre-trial and a Pos-trial Measure in 12 Weeks
Description: change in the number of urgency urinary incontinence episodes as measures by a 3-day voiding diary pre- vs. post-treatment. This includes a baseline measure pre-trial and then a post-trial measure in 12 weeks and then you calculate the difference. The difference between the two measures (baseline vs. post-trial) was then compared with a sample t test.
Time Frame: 3 day voiding diary will be filled out prior to the 12 week PTNS trial and voiding diary will be filled out immediately after the 12 week PTNS trial
Measure: Mean (Standard Deviation); unit: UUI episodes
Arm/Group | Posterior Tibial Nerve Stimulation With Mirabegron | Posterior Tibial Nerve Stimulation Plus Placebo
Number analyzed (Participants) | 20 | 26
UUI episodes | 9.4 (3.9) | 5.3 (5.4)

2. Secondary Outcome: Change in Symptom Distress as Measured by the Urinary Distress Index (UDI-6) Questionnaire Pre- (Baseline Measure) vs. Post-treatment (Post-trial Measure)
Description: This is a quality of life measure using a validated questionnaire called the Urinary Distress Index Scale with a range from 0-100 with higher scores meaning worse urinary distress such as urinary incontinence and leakage and bother with the life stresses related to urinary incontinence. Will include a baseline measure pre-trial and then a post-trial measure (post-trial). This includes a pre-trial measure (baseline) and a post-trial measure and then a calculation of the difference. The difference between the two measures (baseline vs. post-trial) was then compared with a sample t test.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Posterior Tibial Nerve Stimulation With Mirabegron | Posterior Tibial Nerve Stimulation Plus Placebo
Number analyzed (Participants) | 20 | 26
score on a scale | 23.6 (12.9) | 16.3 (14.0)

3. Secondary Outcome: Change in UUI (Urge Urinary Incontinence)/OAB (Overactive Bladder) Quality of Life as Measured by the Incontinence Impact Questionnaire Short Form (IIQ-7) Questionnaire Pre- (Baseline Measure) vs. Post-treatment (Post-trial Measure in 12 Weeks)
Description: The IIQ-7 (Incontinence Impact Questionnaire) is a measure of distress caused by urge urinary incontinence and overactive bladder in the patient. This scale is a scale of 0-100 with 0 being minimal impact and 100 being worse impact and distress. This includes a baseline pre-trial measure and a post-trial measure at 12 weeks. This includes a pre-trial measure (baseline) and then a post-trial measure and then a calculation of the difference. The difference between the two measures (baseline vs. post-trial) was then compared with a sample t test.
Time Frame: pre-trial 0-100 scale measurement and then 12 weeks later post-trial measurement 0-100 with higher scores meaning worse impact.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Posterior Tibial Nerve Stimulation With Mirabegron | Posterior Tibial Nerve Stimulation Plus Placebo
Number analyzed (Participants) | 20 | 26
score on a scale | 29.7 (17.4) | 20.2 (17.6)

4. Secondary Outcome: Change in UUI (Urge Urinary Incontinence)/OAB (Overactive Bladder) Quality of Life as Measured by the Overactive Bladder Questionnaire-Short Form (OAB-q SF) Questionnaire Pre- (Baseline Measure) vs. Post-treatment (Post-trial Measure)
Description: This is the change in Quality of life measure for urge urinary incontinence for the OABq SF scale and it is a 0-100 scale where 0 equals minimum symptoms and 100 equals maximal symptoms. Lower scores indicate better quality of life and higher scores indicate worse quality of life. This includes a pre-trial measure and a post-trial measure at 12 weeks and then a calculation of the difference. The difference between the two measures (baseline vs. post-trial) was then compared with a sample t test.
Time Frame: pre trial measurements as described and then 12 weeks later post-trial measurements as described.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Posterior Tibial Nerve Stimulation With Mirabegron | Posterior Tibial Nerve Stimulation Plus Placebo
Number analyzed (Participants) | 20 | 26
score on a scale | 53.6 (30.0) | 33.3 (35.7)

ADVERSE EVENTS:
Time Frame: During the study, each patient (all 54) were monitored for adverse events from baseline (start of the study) to 12 weeks (the end of the study for each patient.
Description: Adverse events were collected on data sheets at each visit; medication (mirabegron or placebo to match) associated adverse effects such as 1) feeling sick (nausea), 2) constipation, 3) diarrhea, 4) urinary tract infection (UTI), 5) headaches, and 6) feeling dizzy, and for PTNS (posterior tibial nerve stimulation) which included 1) bleeding at the stimulation site, 2) lower extremity swelling, 3) worsening of urinary incontinence, 4) leg cramps, 5) vasovagal response, and 6) generalized headache.
Arm/Group | Posterior Tibial Nerve Stimulation With Mirabegron | Posterior Tibial Nerve Stimulation Plus Placebo
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/27
Other Adverse Events (participants affected / at risk) | 6/27 | 6/27
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Posterior Tibial Nerve Stimulation With Mirabegron (N=27) | Posterior Tibial Nerve Stimulation Plus Placebo (N=27)
Urinary Tract Infection (General disorders) | 3 (3) | 3 (3)
transient leg swelling from PTNS (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-07): https://cdn.clinicaltrials.gov/large-docs/32/NCT04907032/Prot_SAP_001.pdf